CLINICAL TRIAL: NCT02238860
Title: A Randomised Trial Comparing Entacavir and Tenofovir in Patients With HBV Decompensated Cirrhosis
Brief Title: A Trial Comparing Entacavir and Tenofovir in Patients With HBV Decompensated Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad sadik memon, Professor of gastroenterology, Asian Institute Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIMS-hep B-123
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Cirrhosis Due to Hepatitis B
Keywords: Hepatitis B; cirrhosis; Entacavir; enofovir
MeSH Terms: conditions — Hepatitis B; Fibrosis | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entacavir (Active Comparator): Entacavir 0.5 mg (OD) for 48 weeks
  Interventions: Drug: Entacavir; Drug: Tenofovir
- Tenofovir (Active Comparator): Tenofovir 300 mg ,OD for 48 weeks
  Interventions: Drug: Entacavir; Drug: Tenofovir

INTERVENTIONS:
Drug: Entacavir — Entacavir-0.5 mg ,OD,for
  Other Names: ETV
Drug: Tenofovir — Tenofovir ,300 mg,OD,for 48 weeks
  Other Names: TDF or PMPA

SUMMARY:
Entacavir and tenofovir are two first line therapies for chronic hepatitis B. Both agents have been claimed equivalent in treatment, there are no head to head trials available in the literature about there effectiveness in HBV Decompensated Cirrhosis. The investigators aimed to compare safety/efficacy and virological response in patients with HBV Decompensated Cirrhosis.

DETAILED DESCRIPTION:
The effectiveness of entacavir and tenofovir has not been prospectively studied in HBV Decompensated cirrhosis? This prospective, randomised clinical trial will help us in better patient management more efficacy and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age (18 years- 70 years)
* Hbv surface antigen positive > 6 months
* HbeAg (positive or negative both)
* Hbv DNA 10^3
* ALT ULN
* No evidence of HCC
* Platelets count > 30 thousands
* CTP score > 7
* Hepatic encephalopathy (grade 1 - 2 only)
* No prior Drug resistance

Exclusion Criteria:

* Age < 18 years
* HCC patients
* Prior drug resistance
* Current HE > 2
* Solid organ transplantation
* Inadequate hematological function
* Co infection with hepatitis C and HIV
* Autoimmune disorders
* Pregnancy and Breast feeding
* Other hepatic diseases
* Patients on immunosuppressant or chemotherapy agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy | 48 weeks
  EFFICACY ENDPOINTS: EFFICACY ENDPOINTS INCLUDED PLASMA HBV DNA, ALT, HBEAG, HBSAG LOSS AND SEROCONVERION AS WELL AS CTP AND MELD SCORE.

SECONDARY OUTCOMES:
Safety | 48 weeks
  SAFETY ENDPOINTS: SAFETY ANALYSIS INCLUDED CUMALATIVE RATES ON TREATMENT ADVERSE EVENTS, SEREIOUS ADVERSE EFFECTS DISCONTINUATION DUE TO SIDE EFFECTS,DEATH,HCC,RENAL IMPAIRMENT , HEPATIC FLARE AND DEVELOPMENT OF DRUG RESISTANCE.

OTHER OUTCOMES:
Outcome | 48 weeks
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad sadik Memon, Fcps gastro, Principal Investigator — AIMS Institute
Locations (1):
- Asian Institute of medical Sciences, Hyderābād, Sindh, Pakistan